CLINICAL TRIAL: NCT01017692
Title: Variability of Magnetic Resonancy Imaging Interpretation for Lumbar Spinal Stenosis
Brief Title: Magnetic Resonance Imaging (MRI) Interpretations for Lumbar Spinal Stenosis (LSS)
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, William Lavelle, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: 5825-MRI Variability
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2013-09

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumbar Spinal Stenosis: Subjects who have undergone or will undergo an MRI, with symptoms of LSS
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI of lumbar spine for subjects presenting with spinal stenosis symptoms

SUMMARY:
The objective of this study is to establish a relationship between the degree of radiologically established anatomical stenosis and the severity of self-assessed outcome measures in patients that have undergone and MRI.

DETAILED DESCRIPTION:
Magnetic Resonance Imaging(MRI) has become the gold standard of evaluation of lumbar spinal stenosis (LSS. LSS is defined as the narrowing of the spinal canal. Thus far, there has been no formal grading system in literature. Physicians, particularly radiologists, in their interpretations, currently describe the degree of stenosis at each level as normal, mild, moderate or severe. Unfortunately, there is no consensus on criteria of these definitions. Treatments and surgical plans are based primarily on this information. Consequently, the reliability and accuracy of this information is critical in terms of optimizing outcomes.

In this study 50-100 MRI studies of patients diagnosed with symptomatic lumbar spinal stenosis will be collected, de-identified, and assigned a study identification number for tracking purposes. Three "raters" from Upstate and three "rater" from outside the institution, that have experience reviewing MRI's will be asked to review the MRI's and classify the LSS at all lumbar levels as normal, mild, moderate or severe in the central canal, lateral recesses and the neuroforamen. The raters will not have any information about the patients. The MRI's will then be given a new identification number, and the patient's self-assessment questionnaires (which are also de-identified and given the study id number) will be given to the raters, for a second review. The raters will have the patients gender, age and outcomes scores from Short form 36, Visual Analog Scale, Oswestry Disability Index and Zurich Claudication Questionnaires. The raters will classify the MRI, as normal, mild, moderate or severe using the outcomes and information supplied.

The data from both ratings will be compiled and compared to assess the reliability of the radiologically established anatomical stenosis when compared with the subjects outcome scores.

This study is for current patients in Upstate Orthopedics office.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 21 years of age
* Must be able to undergo or have undergone an MRI of the Lumbar spine
* Must be able to read/understand English
* Must be a current patient in our practice

Exclusion Criteria:

* Prisoner

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are seen at SUNY Upstate Medical Univeristy, Department of Orthopedic Surgery office
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
A numeric score will be calculated for the actual percent stenosis at the symptomatic level(s) and will report the predictive power of MRI based on all the analysis of MRI with and without clinical knowledge of patient's presenting symptoms | one year

CONTACTS AND LOCATIONS:
Overall Officials: William F Lavelle, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University-Department of Orthopedics, Syracuse, New York, United States